CLINICAL TRIAL: NCT06625866
Title: Design, Implementation, and Evaluation of Interventions Based on Behavioral Sciences to Reduce Episiotomy Use: a Pilot Study
Brief Title: Evaluation of Interventions Based on Behavioral Sciences to Reduce Episiotomy Use
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Panamericana (Other)
Collaborators: Universidad de la Salud - UNISA (Unknown); IMSS-Bienestar (Unknown); Secretaría de Educación, Ciencia, Tecnología e Innovación de la Ciudad de México (Unknown)
Responsible Party: Principal Investigator, Mario I. Lumbreras-Marquez, MD, MMSc, Professor, Public Health and Epidemiology Department, Universidad Panamericana
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 101 - 101 - 001 - 24
Record Dates: First submitted 2024-09-10; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Episiotomy; Episiotomy Extended by Laceration; Episiotomy Infection; Episiotomy Wound

STUDY DESIGN:
Intervention Model Description: Two hospitals (clusters) will be assigned to intervention and standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Behavioral intervention (Experimental): The healthcare professionals in this hospital will be exposed to behavioral interventions, including feedback and information strategies.
  Interventions: Behavioral: Feedback and information
- Standard of care (No Intervention): The standard of care will be provided in this hospital without exposure to behavioral interventions for healthcare professionals.

INTERVENTIONS:
Behavioral: Feedback and information — The healthcare professionals in the intervention arm will be exposed to feedback and information behavioral strategies. Namely, interns, residents, obstetricians/gynecologists, and nurses will receive written feedback about the episiotomy rates in the hospital each month during the study period. Moreover, at least two academic sessions will be designed to outline the indications, surgical technique, complications, and surgical ethics for the procedure (i.e., episiotomy). Likewise, each session will also include a patient testimonial about their experience during delivery and their follow-up when an episiotomy was performed.
  The feedback intervention will be provided for 2 months, and the feedback intervention + the information intervention will be provided for 2 additional months.
  Arms: Behavioral intervention

SUMMARY:
This pilot study seeks to analyze the impact of interventions based on behavioral economics theory (e.g., feedback and information) on episiotomy use.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare personnel involved in decision-making associated with performing episiotomies who work in the hospital selected to pilot the proposed intervention.

Exclusion Criteria:

* Healthcare personnel who are not involved in the decision-making process over performing episiotomy during delivery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Number of episiotomies performed | During spontaneous or assisted vaginal delivery
  Number of episiotomies performed among patients having a vaginal delivery.
  Episiotomy: surgical incision made in the perineum during childbirth to enlarge the vaginal opening and facilitate the delivery.
  There are two main types of episiotomies, classified based on the direction of the incision: Median (the incision is made straight down from the vaginal opening towards the anus) and mediolateral (the incision is made at an angle [usually 45 degrees] from the vaginal opening towards the side, away from the anus).

SECONDARY OUTCOMES:
Episiotomy indication documented in the medical record | During spontaneous or assisted vaginal delivery
  Number of episiotomies performed with an indication documented in the medical record among patients having a vaginal delivery.
  Potential indications:
  Nonreassuring fetal status, prolonged or difficult labor, operative vaginal delivery, shoulder dystocia, large for gestational age fetus, breech delivery, rigid perineum, maternal fatigue or exhaustion, preterm delivery.
Number of assisted vaginal deliveries | At the time of vaginal delivery
  Number of assisted deliveries among patients having a vaginal delivery. Assisted vaginal delivery refers to the use of specialized instruments, such as forceps or a vacuum device, to help guide the fetal head out of the birth canal during childbirth.
Number of perineal and cervical lacerations (composite outcome) | At the time of spontaneous or assisted vaginal delivery
  Number of perineal and cervical lacerations (composite outcome) among patients having a vaginal delivery.
  The composite outcome will include any of the following:
  Perineal Lacerations:
  First degree: Injury to Perineal skin only. Second degree: Injury to perineum involving perineal muscles but not involving anal sphincter. Third degree: Injury to perineum involving anal sphincter complex. 3a: Less than 50% of external anal sphincter thickness torn. 3b: More than 50% external anal sphincter thickness torn. 3c. Both external anal sphincter and internal sphincter torn. Fourth degree: Injury to perineum involving anal sphincter complex (external anal sphincter and internal anal sphincter) and anal epithelium.
  Cervical Laceration:
  A cervical laceration during delivery refers to a tear or injury to the cervix that occurs during childbirth.
Rate of transfusion of blood products (composite outcome) | Administered in the first 24 hours after delivery
  Administration of any of the following :
  RBCs, fresh frozen plasma (FFP), platelets and cryoprecipitate
Blood loss at the time of delivery | Within the first hour after spontaneous or assisted vaginal delivery
  Estimated or calculated blood loss (mL).
Hematocrit after delivery | Within 24 hours after delivery
  Percentage (%) of red blood cells (RBCs) in the total blood volume.
Pain management after delivery | Administered in the first 24 hours after vaginal delivery
  Description of Nonsteroidal Antiinflammatory Drugs and Opioids administered
Patient satisfaction with the inpatient care received during and after vaginal delivery | Within the first 24 hours after delivery.
  Brief voluntary and anonymous survey designed by the research team to be answered by ~300 patients.
Rate of surgical site infection | In the first 6 weeks after vaginal delivery
  Surgical site infection related to episiotomies, perineal, or cervical lacerations that occurred at the site of these surgical or traumatic wounds after childbirth.
Rate of surgical site dehiscence | In the first 6 weeks after vaginal delivery
  Partial or complete wound reopening along a surgical incision or laceration previously closed (e.g., episiotomies, perineal lacerations, cervical lacerations).
Five-minute Apgar | Neonatal assessment 5 minutes after spontaneous or assisted vaginal delivery
  5-Minute Apgar Score Components:
  The Apgar score assesses five key signs of a newborn's health, each assigned a score of 0, 1, or 2, for a total possible score of 10:
  1. Appearance (skin color)
     * 0: Blue or pale all over.
     * 1: Body pink, but extremities blue.
     * 2: Entire body pink.
  2. Pulse (heart rate)
     * 0: No heartbeat.
     * 1: Fewer than 100 beats per minute.
     * 2: At least 100 beats per minute.
  3. Grimace (reflex irritability, response to stimulation)
     * 0: No response to stimulation.
     * 1: Grimace or weak response when stimulated.
     * 2: Strong cry or active withdrawal in response to stimulation.
  4. Activity (muscle tone)
     * 0: Limp, no movement.
     * 1: Some flexion of extremities.
     * 2: Active movement.
  5. Respiration (breathing effort)
     * 0: Not breathing.
     * 1: Weak or irregular breathing.
     * 2: Strong cry, normal breathing.
Rate of NICU Admission | In the first 24 hours after delivery.
  Transfer and care of a newborn in the Neonatal Intensive Care Unit (NICU) to provide intensive medical care for premature, ill, or high-risk newborns.
Rate of Neonatal death | Within the first 28 days of life
  Neonatal death refers to the death of a newborn within the first 28 days of life. This period is further divided into two phases:
  * Early neonatal death: Neonatal death within the first 7 days of life.
  * Late neonatal death: Neonatal death occurring between 7 and 28 days of life.

IPD SHARING:
Plan to Share IPD: No